CLINICAL TRIAL: NCT04070287
Title: Innovative Tools to Expand HIV Self-Testing
Acronym: I-TEST
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Nigerian Institute of Medical Research (Other Government); University of North Carolina, Chapel Hill (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Juliet Iwelunmor, Professor of Medicine Washington University School of Medicine, Washington University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 30347; 1UG3HD096929-01 (NIH)
Record Dates: First submitted 2019-07-20; First posted 2019-08-28 (Actual); Results first posted 2021-09-14 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: HIV/AIDS; Sexually Transmitted Diseases
Keywords: HIV Prevention; HIV self-testing; young people; Nigeria
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Intervention Pilot
  This study protocol will involve undertaking a prospective one-year assessment of five youth participatory interventions. These interventions are focused on promoting HIV self-testing and referrals to health facilities for other sexually transmitted infections test.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- SMART Pack (Active Comparator): This involves using "SMART Pack" a HIV self-testing kit to promote uptake of HIV self-testing among young people at community centers.
  Interventions: Combination Product: SMART Pack
- Luv Box (Active Comparator): The intervention involves using "Luv Box" a box that include personal hygiene products and HIV self-testing kit as strategy to promote uptake of HIV testing among young people.
  Interventions: Combination Product: Luv Box
- Bili Vibes (Active Comparator): The intervention involves using a program program called "Bili" that leverages community youth events such as football matches as a strategy to promote the uptake of HIV self-testing among young people.
  Interventions: Combination Product: Bili Vibes
- BeterDoc (Active Comparator): This intervention involve using "BeterDoc Safety kits" that includes HIV self-testing kit, location and phone number to the health centers in the community as a strategy to promote update of HIV self-testing among young people.
  Interventions: Combination Product: BeterDoc
- IUNGO (Active Comparator): This intervention involves using a program utilizes community vocational skills training centers to promote uptake of HIV self-testing among young people.
  Interventions: Combination Product: IUNGO

INTERVENTIONS:
Combination Product: SMART Pack — The SMART pack is a re-branded and repackaged box for HIV self-testing kits. The intervention aims to promote distribution of HIVST kits through in institutions, vocational centers, and social media platforms. The intervention would also include a referral systems, where participants provided with the HIV self-testing kits are provided with information with youth-friendly health facilities for uptake of testing for sexually transmitted infections. The intervention would be promoted using flyers at community events and schools. The flyers will provide information on the SMART pack and the location where the pack can be obtained for individuals who are interested. For this pilot study, the intervention will be implemented in Yaba local government area in Lagos state.
  Other Names: The OraQuick®ADVANCERapid HIV-1/2 Antibody Test
  Arms: SMART Pack
Combination Product: Luv Box — The Luv box is packaged in two colors: blue and pink. The LUVBox would be made available in supermarkets, on-line stores, mini-marts, pharmacies, neighborhood stores and markets, for easy accessibility in hard to reach areas. The intervention would be promoted using flyers at community events and schools. The flyers will provide information on the "Luv Box" and the location where the pack can be obtained for individuals who are interested.For this pilot study, the intervention will be implemented in Yaba in Lagos state.
  Other Names: The OraQuick®ADVANCERapid HIV-1/2 Antibody Test
  Arms: Luv Box
Combination Product: Bili Vibes — The HIV self-testing kits will be available for interested individuals at the community youth events. These events and information the HIV self-testing kits will be on flyers that would be promoted at community centers and schools. For this pilot study, the intervention will be implemented in Ngenevu/Bunker communities in Enugu state.
  Other Names: The OraQuick®ADVANCERapid HIV-1/2 Antibody Test
  Arms: Bili Vibes
Combination Product: BeterDoc — The intervention would be promoted using flyers at community events and schools. The flyers will provide information on the "BeterDoc Safety Kits" and the location where the pack can be obtained for individuals who are interested. For this pilot study, the intervention will be implemented in Ibadan, Dugbe and Agbowo in Oyo state.
  Other Names: The OraQuick®ADVANCERapid HIV-1/2 Antibody Test
  Arms: BeterDoc
Combination Product: IUNGO — The intervention would be promoted using flyers at community events and schools. The flyers will provide information on the HIV self-testing kits and the location where the pack can be obtained for individuals who are interested. For this pilot study, the intervention will be implemented in Akure South, Orita-Obele, Ipinsa, Ilara Mokin and Ijare in Ondo state.
  Other Names: The OraQuick®ADVANCERapid HIV-1/2 Antibody Test
  Arms: IUNGO

SUMMARY:
The I-TEST study builds upon two participatory approaches, open challenge contests and entrepreneurship training. The study utilizes open challenge contest to generate youth-driven interventions on strategies to promote HIV self-testing and other testing for other sexually transmitted infections (STIs) among young people in Nigeria. Open challenge contests involves leveraging on the knowledge and strengths of the crowd (in this case young people) to generate solutions to an issue. Following completion of one of the open challenge contest, was the Designathon contest where young people in Nigeria collaborated to develop new services and products for promoting self-testing for HIV and other sexually transmitted diseases, guided by human-centered, design thinking framework. After which, six teams from the Designathon were selected to move onto an Innovation bootcamp. The Innovation bootcamp was a 4-week long accelerated training program for young people to delve into the world of entrepreneurial and innovation management skills, while applying basic research principles. At the end of the course, 5 finalist teams were selected to pilot test their innovation plan in the community for a duration of 6 months, beginning July 2019.

This study is focused on evaluating the effectiveness of these five youth participatory interventions on HIV testing and other key prevention among at risk youth (14-24 years old in Nigeria).This research study will involve undertaking a prospective one-year assessment of these five pilot interventions.

DETAILED DESCRIPTION:
Step 1: Participant enrollment. This will involve recruiting youth to participate in the pilot study. Participant recruitment strategies will include: social media, online, event- and venue based, participant referral, and walk-ins at study clinics. Participant enrollment will be completed by study team.

Step 2: Intervention implementation. Following participant recruitment and enrollment in the study. Study participants will be assigned to one of the 5 youth participatory interventions focused on expanding the uptake of HIV self-testing and key HIV prevention services. The pilot intervention implementation would occur for 6 months. Nigerian Institute of Medical Research (NMIR) will provide local training on HIV prevention to the five participatory interventions following their existing guidelines.The participatory interventions will be conducted in the locations of the five teams who emerged as winners from the innovation boot-camp. These participatory interventions will only provide HIV self-testing kits and instructions of how to perform the test to participants. They will also provide referral coupons to youth friendly centers for sexually transmitted infections (STI) screening and treatment and pre-exposure prophylaxis (PrEP) awareness and initiation for at-risk youth. The referral coupons are intended to provide study participants information on trained youth friendly centers that are involved with the research. The referral coupons give the study participants access to other sexually transmitted infections (STI) screening and treatment and pre-exposure prophylaxis (PrEP) awareness and initiation at these health facilities. The intervention only provide participants with the HIV self-testing kits and then refer them to youth-friendly health facilities for other testing services. The intervention does not involve monitoring HIV self-testing procedure, the investigators will only be asking for self-reported HIV testing and other sexually transmitted diseases testing.

Step 3: Baseline data collection. After allocation of participants into the intervention, study team will collect baseline data on HIV testing history, sexual behavior history, youth participation experience, and other related outcomes will be collected (survey questionnaire attached) from recruited participants. Participants mobile phone numbers will also be collected as tracking information for follow-up and retention in a coupon format. The mobile phone numbers would be used to contact study participants through text messages and phone calls. These contacts would serve as reminders for participants to participate in follow-up data collection. The mobile phone service charge would be covered by the research. No other personal identifiers will be collected and no biological specimens will be collected at baseline. The investigators will obtain informed consent before proceeding with any data collection.

Step 4:Health facilities training. For the purposes of this research study, the Nigerian Institute of Medical Research team would provide training to youth-friendly health centers currently working with the Nigerian Institute of Medical Research based on the World Health Organization guidebook for youth-friendly health services (handbook is attached).The training would be to ensure that these health facilities are trained to provide youth friendly services to participants who be referred to receive STI screening, STI treatment and PrEP awareness and initiation. Following the training, the NIMR research team would in charge of collecting data to record record participants HIV self-testing uptake as well as uptake of STI screening, STI treatment and PrEP awareness and initiation.

Step 5: Follow up surveys at 3 and 6 months: At 3 and 6 months post intervention implementation, study team will collect similar baseline data from study participants. The follow-up survey will assess HIV testing, sexual behavior history, youth participation experience and other related outcomes will be collected (survey questionnaire attached) from recruited participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14-24
2. Self-reported HIV negative or unknown HIV status
3. Current resident of Lagos, Ondo, Oyo, and Enugu with plans to stay in city for the next 6 months
4. Able to complete survey in English (the national language of Nigeria)
5. All participants must agree to an informed consent and provide their cell mobile number for follow-up and retention

Exclusion Criteria:

1. Younger than 14 and older than 24
2. Inability to comply with study protocol
3. Illness, cognitive impairment or threatening behavior with acute risk to self or others
4. No informed consent
5. No contact phone number
6. Do not reside in Lagos, Ondo, Oyo, and Enugu

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 388 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Iwelunmor, PhD, Principal Investigator — Washington University School of Medicine; Joseph Tucker, MD, Principal Investigator — University of North Carolina, Chapel Hill; Oliver Ezechi, MD, Principal Investigator — Nigerian Institute of Medical Research
Locations (1):
- Nigerian Institute of Medical Research, Yaba, Lagos, Nigeria

REFERENCES:
- [Background] Nigeria Framework. National HIV and AIDS Strategic Framework. 2017-2021.
- [Background] NACA. Federal Republic of Nigeria, Global AIDS Report: Country Progress Report. 2015. Accessed Novembner, 2015.
- [Background] NDHS. National Population Commision; Nigerian Demographic and Health Survey Reports. 2013.
- [Background] Asaolu IO, Gunn JK, Center KE, Koss MP, Iwelunmor JI, Ehiri JE. Predictors of HIV Testing among Youth in Sub-Saharan Africa: A Cross-Sectional Study. PLoS One. 2016 Oct 5;11(10):e0164052. doi: 10.1371/journal.pone.0164052. eCollection 2016. PMID 27706252
- [Background] Sekoni AO, Somefun EO, Fatoba OO, Onajole AT. Use of HIV Screening Services and Sexual Behavior of In-School Adolescents in Surulere LGA, Lagos State. Nig Q J Hosp Med. 2015 Jul-Sep;25(3):202-8. PMID 27295814
- [Background] Sam-Agudu NA, Folayan MO, Ezeanolue EE. Seeking wider access to HIV testing for adolescents in sub-Saharan Africa. Pediatr Res. 2016 Jun;79(6):838-45. doi: 10.1038/pr.2016.28. Epub 2016 Feb 16. PMID 26882367
- [Background] Tucker JD, Wei C, Pendse R, Lo YR. HIV self-testing among key populations: an implementation science approach to evaluating self-testing. J Virus Erad. 2015 Jan;1(1):38-42. doi: 10.1016/S2055-6640(20)31145-6. PMID 26005717
- [Background] Indravudh PP, Sibanda EL, d'Elbee M, Kumwenda MK, Ringwald B, Maringwa G, Simwinga M, Nyirenda LJ, Johnson CC, Hatzold K, Terris-Prestholt F, Taegtmeyer M. 'I will choose when to test, where I want to test': investigating young people's preferences for HIV self-testing in Malawi and Zimbabwe. AIDS. 2017 Jul 1;31 Suppl 3(Suppl 3):S203-S212. doi: 10.1097/QAD.0000000000001516. PMID 28665878
- [Background] Smith P, Wallace M, Bekker LG. Adolescents' experience of a rapid HIV self-testing device in youth-friendly clinic settings in Cape Town South Africa: a cross-sectional community based usability study. J Int AIDS Soc. 2016 Jan;19(1):21111. doi: 10.7448/IAS.19.1.21111. Epub 2016 Dec 23. PMID 28406597
- [Background] Jennings L, Conserve DF, Merrill J, Kajula L, Iwelunmor J, Linnemayr S, Maman S. Perceived Cost Advantages and Disadvantages of Purchasing HIV Self-Testing Kits among Urban Tanzanian Men: An Inductive Content Analysis. J AIDS Clin Res. 2017 Aug;8(8):725. doi: 10.4172/2155-6113.1000725. Epub 2017 Aug 31. PMID 29051841
- [Background] WHO. HIV Testing Services: WHO recommends HIV Self-testing. Geneva2016.
- [Background] Ozer EJ. Youth-Led Participatory Action Research: Developmental and Equity Perspectives. Adv Child Dev Behav. 2016;50:189-207. doi: 10.1016/bs.acdb.2015.11.006. Epub 2016 Jan 25. PMID 26956074
- [Background] Ozer EJ, Piatt AA, Holsen I, Larsen T, Lester J, Ozer EM. INNOVATIVE APPROACHES TO PROMOTING POSITIVE YOUTH DEVELOPMENT IN DIVERSE CONTEXTS. Positive Youth Development in Global Contexts of Social and Economic Change. 2016:12.
- [Background] Ozer EJ. Youth-led participatory action research. Handbook of methodological approaches to community-based research: Qualitative, quantitative, and mixed methods. 2016:263-272. 15.Cammarota J, Fine M. Revolutionizing education : youth participatory action research in motion. New York, NY: Routledge; 2008.
- [Background] Cammarota J, Fine M. Revolutionizing education : youth participatory action research in motion. New York, NY: Routledge; 2008.
- [Background] Ozer EJ, Newlan S, Douglas L, Hubbard E. "Bounded" empowerment: analyzing tensions in the practice of youth-led participatory research in urban public schools. Am J Community Psychol. 2013 Sep;52(1-2):13-26. doi: 10.1007/s10464-013-9573-7. PMID 23444005
- [Background] Jacquez F, Vaughn LM, Wagner E. Youth as partners, participants or passive recipients: a review of children and adolescents in community-based participatory research (CBPR). Am J Community Psychol. 2013 Mar;51(1-2):176-89. doi: 10.1007/s10464-012-9533-7. PMID 22718087
- [Background] Zhang Y, Kim JA, Liu F, Tso LS, Tang W, Wei C, Bayus BL, Tucker JD. Creative Contributory Contests to Spur Innovation in Sexual Health: 2 Cases and a Guide for Implementation. Sex Transm Dis. 2015 Nov;42(11):625-8. doi: 10.1097/OLQ.0000000000000349. PMID 26462186
- [Background] Halpern R. The means to grow up: Reinventing apprenticeship as a developmental support in adolescence. Routledge; 2013.
- [Background] Louw J, Peltzer K, Chirinda W. Correlates of HIV risk reduction self-efficacy among youth in South Africa. ScientificWorldJournal. 2012;2012:817315. doi: 10.1100/2012/817315. Epub 2012 Nov 28. PMID 23251106
- [Background] Sayles JN, Pettifor A, Wong MD, MacPhail C, Lee SJ, Hendriksen E, Rees HV, Coates T. Factors associated with self-efficacy for condom use and sexual negotiation among South african youth. J Acquir Immune Defic Syndr. 2006 Oct 1;43(2):226-33. doi: 10.1097/01.qai.0000230527.17459.5c. PMID 16951647
- [Background] Tiffany JS, Exner-Cortens D, Eckenrode J. A New Measure for Assessing Youth Program Participation. J Community Psychol. 2012 Apr 1;40(3):277-291. doi: 10.1002/jcop.20508. PMID 23843679
- [Derived] Gbaja-Biamila T, Obiezu-Umeh C, Nwaozuru U, Rosenberg NE, Igbokwe M, Oladele D, Musa AZ, Idigbe I, Conserve D, Day S, Tahlil K, Ong J, Muessig K, Nkengasong S, Xian H, Tucker JD, Ezechi O, Iwelunmor J. Awareness of, willingness to use, and experiences with Pre-exposure prophylaxis among youth in Nigeria. BMC Health Serv Res. 2024 Sep 27;24(1):1128. doi: 10.1186/s12913-024-11459-1. PMID 39334111

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred through a combination of community-based events, social media platforms, and peer referral.
Period: Overall Study
Arm/Group | SMART Pack | Luv Box | Bili Vibes | BeterDoc | IUNGO
Started (Youth (aged 14-24 years) enrolled in the study) | 114 | 86 | 81 | 11 | 96
Completed (Youth retained through a 6-month follow-up period) | 103 | 44 | 75 | 7 | 95
Not Completed | 11 | 42 | 6 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SMART Pack | Luv Box | Bili Vibes | BeterDoc | IUNGO | Total
Number analyzed (Participants) | 114 | 86 | 81 | 11 | 96 | 388
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.0 (2.8) | 21.3 (2.3) | 21.1 (1.5) | 20.7 (2.1) | 21.1 (2.1) | 21.1 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 40 | 30 | 4 | 32 | 160
  Male | 60 | 46 | 51 | 7 | 64 | 228
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Yoruba | 49 | 57 | 0 | 10 | 71 | 187
  Igbo | 30 | 20 | 70 | 0 | 10 | 130
  Other ethnicity (i.e. Hausa/Fulani) | 35 | 9 | 7 | 1 | 14 | 66
  Missing | 0 | 0 | 4 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Uptake of HIV Self-testing Over the 3 Months Follow-up
Description: Proportion of participants who reported to have self-tested for HIV at 3-month after baseline.
Time Frame: 3 months following the first encounter
Measure: Count of Participants; unit: Participants
Arm/Group | SMART Pack | Luv Box | Bili Vibes | BeterDoc | IUNGO
Number analyzed (Participants) | 114 | 86 | 81 | 11 | 96
Participants | 19 | 7 | 24 | 4 | 22
Statistical Analysis 1: Comparison: SMART Pack vs Luv Box vs Bili Vibes vs BeterDoc vs IUNGO; Test type: Superiority; p < 0.05, Chi-squared

2. Secondary Outcome: Uptake of HIV Testing Over the 6 Months Follow-up
Description: Proportion of participants who reported to have self-tested for HIV at 6-month after baseline.
Time Frame: 6-month
Measure: Count of Participants; unit: Participants
Arm/Group | SMART Pack | Luv Box | Bili Vibes | BeterDoc | IUNGO
Number analyzed (Participants) | 114 | 86 | 81 | 11 | 96
Participants | 98 | 32 | 64 | 4 | 91
Statistical Analysis 1: Comparison: SMART Pack vs Luv Box vs Bili Vibes vs BeterDoc vs IUNGO; Test type: Superiority; p < 0.05, Chi-squared

3. Secondary Outcome: Uptake of Syphilis Testing
Description: Proportion of participants who reported syphilis testing at baseline and 6-month.
Time Frame: 6-month
Measure: Count of Participants; unit: Participants
Arm/Group | SMART Pack | Luv Box | Bili Vibes | BeterDoc | IUNGO
Number analyzed (Participants) | 114 | 86 | 81 | 11 | 96
Participants
  Baseline | 3 | 4 | 8 | 0 | 3
  6-month | 47 | 5 | 25 | 0 | 73
Statistical Analysis 1: Comparison: SMART Pack vs Luv Box vs Bili Vibes vs BeterDoc vs IUNGO; Test type: Superiority; p < 0.05, Chi-squared

4. Secondary Outcome: Uptake of Gonorrhea Testing
Description: Proportion of participants who reported gonorrhea testing at baseline and 6-month.
Time Frame: 6-month
Measure: Count of Participants; unit: Participants
Arm/Group | SMART Pack | Luv Box | Bili Vibes | BeterDoc | IUNGO
Number analyzed (Participants) | 114 | 86 | 81 | 11 | 96
Participants
  Baseline | 5 | 5 | 3 | 0 | 5
  6-month | 46 | 2 | 23 | 0 | 64
Statistical Analysis 1: Comparison: SMART Pack vs Luv Box vs Bili Vibes vs BeterDoc vs IUNGO; Test type: Superiority; p < 0.05, Chi-squared

5. Secondary Outcome: Uptake of Hepatitis b Testing
Description: Proportion of participants who reported hepatitis B testing.
Time Frame: 6-month
Measure: Count of Participants; unit: Participants
Arm/Group | SMART Pack | Luv Box | Bili Vibes | BeterDoc | IUNGO
Number analyzed (Participants) | 114 | 86 | 81 | 11 | 96
Participants
  Baseline | 3 | 8 | 31 | 3 | 8
  6-month | 46 | 6 | 45 | 2 | 75
Statistical Analysis 1: Comparison: SMART Pack vs Luv Box vs Bili Vibes vs BeterDoc vs IUNGO; Test type: Superiority; p < 0.05, Chi-squared

6. Secondary Outcome: Uptake of Chlamydia Testing
Description: Proportion of participants who reported chlamydia testing at baseline and 6-month.
Time Frame: 6-month
Measure: Count of Participants; unit: Participants
Arm/Group | SMART Pack | Luv Box | Bili Vibes | BeterDoc | IUNGO
Number analyzed (Participants) | 114 | 86 | 81 | 11 | 96
Participants
  Baseline | 1 | 3 | 1 | 0 | 0
  6-month | 45 | 3 | 21 | 0 | 73
Statistical Analysis 1: Comparison: SMART Pack vs Luv Box vs Bili Vibes vs BeterDoc vs IUNGO; Test type: Superiority; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | SMART Pack | Luv Box | Bili Vibes | BeterDoc | IUNGO
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/86 | 0/81 | 0/11 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/86 | 0/81 | 0/11 | 0/96
Other Adverse Events (participants affected / at risk) | 0/114 | 0/86 | 0/81 | 0/11 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT04070287/Prot_SAP_001.pdf
  • Informed Consent Form (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT04070287/ICF_000.pdf